CLINICAL TRIAL: NCT03344549
Title: Effect of Nutritional Intervention Through Teleconsultation on Glomerular Filtration Rate and Glycated Hemoglobin A1c in Patients With Diabetic Kidney Disease in Stage G3a, G3b and G4.
Brief Title: Effect of the Teleconsultation of Renal Nutrition on Renal Function and Glycemic Control in Patients With DKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil Juan I. Menchaca (Other)
Responsible Party: Principal Investigator, Andrea Garcia Contreras, Ari Cisneros Hernández, Hospital Civil Juan I. Menchaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCN001
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2022-10

CONDITIONS: Diet Modification; Diabetic Kidney Disease; Chronic Kidney Diseases
Keywords: eHealth; Nutrition Therapy; Telehealth; Diabetic Kidney Disease; Chronic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: In the experimental group, the nutritional intervention will be done through teleconsultation with the free technological tool chosen (the patients from home and the nutritionist from the remote clinic); and in the control group will be offered the nutritional intervention through face-to-face consultations carried out by the nutritionist of the nutrition service of the institution, both arms will be intervened monthly for four months, the duration of the sessions will be 45 minutes and will include evaluation or re-evaluation of dietary data, diagnosis, treatment and educational approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleconsultation (Experimental): In the patients of the experimental group, the nutritional intervention is carried out through teleconsultation with the free technological tool chosen (the patients from home and the nutritionist from the remote clinic).
  Interventions: Behavioral: Renal nutrition teleconsultation
- Face-to-face consultation (Other): In the patients of the other group, the nutritional intervention is offered through face-to-face consultations carried out by the nutritionist of the nutrition service of the institution.
  Interventions: Behavioral: Face-to-face consultation of renal nutrition

INTERVENTIONS:
Behavioral: Renal nutrition teleconsultation — Renal Nutritional teleconsultation for patients with diabetic kidney disease without dialysis, monthly for 4 months.
  Arms: Teleconsultation
Behavioral: Face-to-face consultation of renal nutrition — Face-to-face consultation of renal nutrition for patients with diabetic kidney disease without dialysis, monthly for 4 months.
  Arms: Face-to-face consultation

SUMMARY:
The modern era is characterized by progress, development and social and economic globalization. Currently the electronic technology has applications in a wide variety of work areas. A clear example of this, is telemedicine. The technological tools are increasingly used every day in the improvement of the processes and the attention in health, in the last decades, telemedicine has grown exponentially becoming more accessible to the population.

On the other hand, and in the same way, the number of people with chronic degenerative diseases such as diabetes and chronic kidney disease are increasing with alarming numbers, The health system can not offer the attention to the great demand. The strategies used until now for its management have gradually evolved towards a more effective prevention and treatment approach which requires a multidisciplinary team. Investigate the use of new tools that promise to improve the service, has also become a prevailing need. Therefore, the purpose of this study is to know the effect of nutritional teleconsultation on renal function and glycemic control of patients with Diabetic Kidney Disease (DKD) in pre-dialysis stages (specifically G3a, G3b and G4).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is the result of various chronic-degenerative diseases, including diabetes mellitus. In Mexico, it is considered a catastrophic disease due to the increasing number of cases, high investment costs and human resources, limited infrastructure, late detection of the disease, and high rates of morbidity and mortality in substitution programs.

So far, there is no record of patients with CKD in Mexico, so the precise number of patients in any of their stages is unknown. International databases, estimate an incidence of 421 patients with terminal CKD treated per million of population per year in our country (represented by the state of Jalisco), and a prevalence of 1,568 cases per million of population; figures that are considered the highest in the world.

Currently our country lives an extraordinarily complex scenario, has shown the highest rate of incidence of terminal kidney disease in recent years, which may be related, at least in part, to the increase in the prevalence of risk factors and the incongruence between needs of patients and the health care system, largely designed for the management of acute diseases. The CKD is among the first 10 causes of general mortality in Mexico, with a survival calculated in average months, from the entrance to a substitution therapy, of 30.6 months. The medical expense provided by the Mexican Institute of Social Security (an public agency that provides coverage to 66% of Mexicans with social security), for the treatment of terminal CKD in 2007, was estimated at $ 4 billion pesos, equivalent 60% of the total medical expense; and it is estimated that, due to the high incidence rates, in 2043 the investment costs will reach 20 billion pesos, figures that can not be paid.

The dimensions of chronic kidney disease show it as a public health problem that requires the creation of new intervention and education programs focused on the prevention of kidney disease and its causes. Currently, doctors have serious difficulties in providing optimal management. It is common for patients during the early stages of CKD not to comply with recommendations for effective control. They usually present negative life habits, difficult to change only with medical intervention. Many of the risk factors for both the onset and progression of CKD are related to unhealthy eating habits. It is widely known that, optimizing the quality of diet and lifestyles, in individuals with CKD at early stages have substantial benefits in terms of preventing the incidence and progression of the disease, as well as in the mortality of this population. Interventions based on multidisciplinary models, developed in populations at risk and in early stages of kidney disease have proven useful for delaying progression and postponing patients' admission to substitution therapy.

As the CKD progresses, the risk of presenting complications such as malnutrition, hyperphosphatemia and hyperkalemia increases significantly, which increases the risk of morbidity and mortality, especially in more advanced stages of the disease. Nutrition interventions to control and modify these risk behaviors become key points for the management of patients with CKD.

A better CKD care also requires economic resources, needs a greater number of nephrologists, nutritionists, nurses and other health professionals specialized in this disease entity. In Mexico, there are only 750 certified specialists in nephrology, the nephrologist patient ratio is 1: 204, values below the demand for health services. A similar analysis carried out in nutrition professionals in our country indicates that, in 2012, there were 2.4 nutritionists per 1,000 inhabitants, of whom only 78% worked in nutrition-related activities. In addition, the area of renal nutrition is little explored by health professionals, due to the lack of specialty certifications, the few existing courses lose rigor and formality due to the lack of an organ that regulates them; all this results in limited access to quality health care.

Deficiencies in the function and structure of health programs for chronic diseases prevent the achievement of good results; and in addition to this, when adherence to treatment is tested, only 44% of patients manage to maintain an adequate adherence that improves prognosis and modifies the natural course of the disease. Studies reveal that patients with chronic kidney disease are often dissatisfied with the communication they have with their health care provider and perceive little or no knowledge about their diagnosis and treatment. Some of the external agents that exacerbate this scenario in Mexico are: social inequality, difficult access to health institutions, the educational level of the population and the economy of the country. In contrast to this and as part of a possible solution, globalization has allowed, as the technology develops, to provide users with access to a wide variety of applications and health portals. According to the National Survey of Availability and Use of Information Technologies in Households in México, 57.4% of the population in Mexico call themselves Internet users and 71.5% as mobile phone users, of which 70.7% declare surfing in Internet through your mobile device. Currently with the internet there is a great variety of information for the patient with CKD, which offers facilities in the understanding of the disease.

Telemedicine emerged with the aim of allowing the health professional to meet the patient when it was otherwise impossible; However, today health providers also use mobile technology to connect with their patients and thus improve their overall relationship, strengthen the patient's autonomy and their ability to face everyday health problems and be more active in their own caring, all these skills suitable for the optimal care of the population with CKD.

Telemedicine in the nephrology has been used to improve different processes, shown that it reduces the waiting times for consultation with the specialist, decreases the number of patients who are referred to the nephrologist without being necessary, decreases costs and increases the coverage area of the service provider. Although there are studies that do not find the superiority in the effectiveness of synchronous telemedicine compared with conventional intervention, others conclude that effectiveness is similar, with the great benefit in reducing costs for transfer and / or for absence from work, which exposes synchronous telemedicine as an available and safe option for clinical practice.

There are few studies of telemedicine that offer specialized nutritional intervention through teleconsultations, the most developed in patients with diabetes mellitus with inconclusive results, however, none (as far as we have knowledge) in patients with CKD. Therefore, the interest of knowing the effect of the nutrition teleconsultation on renal function and glycemic control in the patient with diabetic kidney disease in stages G3a, G3b and G4 was born.

The working hypothesis is that, there is a difference between the nutritional intervention through teleconsultation and the face-to-face consultation in patients with diabetic kidney disease in stage G3a, G3b and G4.

For the calculation of sample size, the formula was used to compare means of independent samples. A size of 34 patients per group was estimated, considering an expected difference in the estimated glomerular filtration rate of 5.82 ml / min / 1.73 m2 reported in a previous study.

The nutritional intervention was considered as the independent variable, which consists of providing nutritional therapy through two modalities, face-to-face consultations in the hospital or through teleconsultations, with a monthly frequency for 4 months. The duration of each consultation is approximately 45 minutes and includes the evaluation or re-evaluation, diagnosis, treatment and educational approach. It will be measured as assistance or non-attendance to the consultation. Non-attendance to more than two consultations is considered an exclusion criterion for the subject.

Two dependent variables were considered, the glycated hemoglobin (HbA1c), which is defined as the result obtained in percentage (%) of the blood glycated hemoglobin test. And the estimated glomerular filtration rate (eGFR), which is defined as the result obtained in milliliters per minute per 1.73 square meters of body area (thousand ml / min / 1.73m2), based on the calculation of the mathematical formula proposed by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) for the estimation of the glomerular filtration rate.

PROCESS

The detection of patients is carried out in the nephrology department of the Juan I. Menchaca hospital, both in the morning and afternoon sessions. The identification of patients is carried out during the consultation with the nephrologist, where the selection criteria are evaluated and the patient is invited to participate in the study and to sign the agree consent.

After the patient's acceptance to participate in the study, the initial evaluation is carried out, which includes contact, demographic, anthropometric and dietary data; and the patient is trained to fill the dietary record at home. Anthropometric data are evaluated by standardized nutritionist trained with the correct technique. The biochemical indicators are requested by the nephrologist at the time of the consultation and the results of these are obtained from the institution's own data system.

After the initial evaluation, the probabilistic group assignment is carried out with the simple method without replacement, which is carried out using a sealed envelope. After the appointment of the group, the patient is scheduled for his first nutrition consultation (both arms).

In the teleconsultation group, two days before the first nutrition consultation, the patient is advised by telephone - or the family member in charge - about the use of the free technological tool to be used during the video conference.

In the patients of the intervention group, the nutritional intervention is carried out through teleconsultation with the free technological tool chosen (the patients from home and the nutritionist from the remote clinic); and the patients of the control group are offered the nutritional intervention through face-to-face consultations carried out by the nutritionist of the nutrition service of the institution. All patients will be confirmed by phone the date and time of their next nutrition consultation, both the control group and the intervention group.

The evaluation of the glycated hemoglobin (HbA1c) and the estimated glomerular filtration rate (eGFR), will be done at the beginning and at the end of the intervention. Adherence is also evaluated at the beginning and end, by means of dietary records for the calculation of energy and protein intake.

STATISTIC ANALYSIS For the comparison of proportions between the groups, it will be done with X2 or Fisher's exact test and to compare quantitative variables, Student's T or Mann-Whitney U will be used. For the intra-group comparisons, Mc Nemar will be used for the qualitative variables and Anova for repeated samples or Friedman's Anova for the quantitative variables. For the analysis of the interaction or intervening variables, a stratified statistical analysis will be carried out, using contingency tables and the Mantel-Haenszel method. The results will be considered statistically significant if the value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic kidney with eGFR <60 ml / min / 1.73m2 and ≥15 ml / min / 1.73m2, (stage G3a, G3b and G4 respectively).
* Patients who can read and write.
* Patients who have access to the internet and have a computer, tablet or smartphone.
* Patients who signed the voluntary agreement to participate.

Exclusion Criteria:

* Patients who have received prior nutritional treatment for the control of diabetic kidney disease.
* Patients with actual consumption of food supplements and / or keto analogues.
* Patients with anemia or recent transfusions (in the last 3 months).
* Patients with serious complications (chronic infection, septicemia, cancer, HIV, Alzheimer's, uncontrolled heart failure, liver failure, etc.).
* Patients with serious difficulties in communication or intellectual deficit that impedes the ability to understand the intervention.
* Patients with refractory arterial hypertension.
* Patients who do not attend ≥ 2 nutritional interventions.
* Patients who present serious complications during the intervention (chronic infection, septicemia, cancer, HIV, Alzheimer's, uncontrolled heart failure, liver failure, etc.).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Cisneros, Bachelor, Principal Investigator — Hospital Civil Juan I. Menchaca
Locations (1):
- Hospital Civil Nuevo Juan I Menchaca, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Garcia G, Marquez-Magana I, Renoirte-Lopez K, Perez-Cortes G, Salazar Gutierrez ML, Klarenbach S, Lloyd A, Tonelli M. Screening for kidney disease on World Kidney Day in Jalisco, Mexico. J Nephrol. 2010 Mar-Apr;23(2):224-30. PMID 20119929
- [Background] Martinez-Ramirez HR, Cortes-Sanabria L, Rojas-Campos E, Hernandez-Herrera A, Cueto-Manzano AM. Multidisciplinary strategies in the management of early chronic kidney disease. Arch Med Res. 2013 Nov;44(8):611-5. doi: 10.1016/j.arcmed.2013.10.013. Epub 2013 Nov 8. PMID 24215785
- [Background] Obrador GT, Garcia-Garcia G, Villa AR, Rubilar X, Olvera N, Ferreira E, Virgen M, Gutierrez-Padilla JA, Plascencia-Alonso M, Mendoza-Garcia M, Plascencia-Perez S. Prevalence of chronic kidney disease in the Kidney Early Evaluation Program (KEEP) Mexico and comparison with KEEP US. Kidney Int Suppl. 2010 Mar;(116):S2-8. doi: 10.1038/ki.2009.540. PMID 20186176
- [Background] Paniagua R, Ramos A, Fabian R, Lagunas J, Amato D. Chronic kidney disease and dialysis in Mexico. Perit Dial Int. 2007 Jul-Aug;27(4):405-9. PMID 17602147
- [Background] Dunkler D, Kohl M, Teo KK, Heinze G, Dehghan M, Clase CM, Gao P, Yusuf S, Mann JF, Oberbauer R. Dietary risk factors for incidence or progression of chronic kidney disease in individuals with type 2 diabetes in the European Union. Nephrol Dial Transplant. 2015 Aug;30 Suppl 4:iv76-85. doi: 10.1093/ndt/gfv086. PMID 26209742
- [Background] Diaz-Lopez A, Babio N, Martinez-Gonzalez MA, Corella D, Amor AJ, Fito M, Estruch R, Aros F, Gomez-Gracia E, Fiol M, Lapetra J, Serra-Majem L, Basora J, Basterra-Gortari FJ, Zanon-Moreno V, Munoz MA, Salas-Salvado J; PREDIMED Study Investigators. Mediterranean Diet, Retinopathy, Nephropathy, and Microvascular Diabetes Complications: A Post Hoc Analysis of a Randomized Trial. Diabetes Care. 2015 Nov;38(11):2134-41. doi: 10.2337/dc15-1117. Epub 2015 Sep 13. PMID 26370380
- [Background] Foster MC, Hwang SJ, Massaro JM, Jacques PF, Fox CS, Chu AY. Lifestyle factors and indices of kidney function in the Framingham Heart Study. Am J Nephrol. 2015;41(4-5):267-74. doi: 10.1159/000430868. Epub 2015 May 20. PMID 25998023
- [Background] Pisani A, Riccio E, Bellizzi V, Caputo DL, Mozzillo G, Amato M, Andreucci M, Cianciaruso B, Sabbatini M. 6-tips diet: a simplified dietary approach in patients with chronic renal disease. A clinical randomized trial. Clin Exp Nephrol. 2016 Jun;20(3):433-42. doi: 10.1007/s10157-015-1172-5. Epub 2015 Oct 9. PMID 26453483
- [Background] Wright Nunes JA, Wallston KA, Eden SK, Shintani AK, Ikizler TA, Cavanaugh KL. Associations among perceived and objective disease knowledge and satisfaction with physician communication in patients with chronic kidney disease. Kidney Int. 2011 Dec;80(12):1344-51. doi: 10.1038/ki.2011.240. Epub 2011 Aug 10. PMID 21832984
- [Background] Diamantidis CJ, Becker S. Health information technology (IT) to improve the care of patients with chronic kidney disease (CKD). BMC Nephrol. 2014 Jan 9;15:7. doi: 10.1186/1471-2369-15-7. PMID 24405907
- [Background] Russo JE, McCool RR, Davies L. VA Telemedicine: An Analysis of Cost and Time Savings. Telemed J E Health. 2016 Mar;22(3):209-15. doi: 10.1089/tmj.2015.0055. Epub 2015 Aug 25. PMID 26305666
- [Background] Scherpbier-de Haan ND, van Gelder VA, Van Weel C, Vervoort GM, Wetzels JF, de Grauw WJ. Initial implementation of a web-based consultation process for patients with chronic kidney disease. Ann Fam Med. 2013 Mar-Apr;11(2):151-6. doi: 10.1370/afm.1494. PMID 23508602
- [Background] Fernandes NM, Bastos MG, Oliveira NA, Costa Ado V, Bernardino HS. Telemedicine: Development of a distance care system for pre-dialysis chronic kidney disease patients. J Bras Nefrol. 2015 Jul-Sep;37(3):349-58. doi: 10.5935/0101-2800.20150055. English, Portuguese. PMID 26398645
- [Background] Su D, McBride C, Zhou J, Kelley MS. Does nutritional counseling in telemedicine improve treatment outcomes for diabetes? A systematic review and meta-analysis of results from 92 studies. J Telemed Telecare. 2016 Sep;22(6):333-47. doi: 10.1177/1357633X15608297. Epub 2015 Oct 6. PMID 26442959
- [Background] Ishani A, Christopher J, Palmer D, Otterness S, Clothier B, Nugent S, Nelson D, Rosenberg ME; Center for Innovative Kidney Care. Telehealth by an Interprofessional Team in Patients With CKD: A Randomized Controlled Trial. Am J Kidney Dis. 2016 Jul;68(1):41-9. doi: 10.1053/j.ajkd.2016.01.018. Epub 2016 Mar 2. PMID 26947216
- [Background] Kelly JT, Reidlinger DP, Hoffmann TC, Campbell KL. Telehealth methods to deliver multifactorial dietary interventions in adults with chronic disease: a systematic review protocol. Syst Rev. 2015 Dec 22;4:185. doi: 10.1186/s13643-015-0170-8. PMID 26693940
- [Background] Rasmussen OW, Lauszus FF, Loekke M. Telemedicine compared with standard care in type 2 diabetes mellitus: A randomized trial in an outpatient clinic. J Telemed Telecare. 2016 Sep;22(6):363-8. doi: 10.1177/1357633X15608984. Epub 2015 Oct 14. PMID 26468213
- [Background] Izquierdo R, Lagua CT, Meyer S, Ploutz-Snyder RJ, Palmas W, Eimicke JP, Kong J, Teresi JA, Shea S, Weinstock RS. Telemedicine intervention effects on waist circumference and body mass index in the IDEATel project. Diabetes Technol Ther. 2010 Mar;12(3):213-20. doi: 10.1089/dia.2009.0102. PMID 20151772
- [Background] Bashshur RL, Shannon GW, Smith BR, Woodward MA. The empirical evidence for the telemedicine intervention in diabetes management. Telemed J E Health. 2015 May;21(5):321-54. doi: 10.1089/tmj.2015.0029. Epub 2015 Mar 25. PMID 25806910
- [Background] Desroches S, Lapointe A, Ratte S, Gravel K, Legare F, Turcotte S. Interventions to enhance adherence to dietary advice for preventing and managing chronic diseases in adults. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD008722. doi: 10.1002/14651858.CD008722.pub2. PMID 23450587
- See also: National Survey of Occupation and Employment, 2016 — http://www3.inegi.org.mx/sistemas/temas/default.aspx?s=est&c=25433&t=1.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Teleconsultation | Face-to-face Consultation
Started | 26 | 27
Completed | 19 | 12
Not Completed | 7 | 15
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Dialysis | 2 | 0
Not completed — Cancer | 1 | 0
Not completed — Lack of electronic device | 1 | 0
Not completed — Transportation difficulty | 0 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teleconsultation | Face-to-face Consultation | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.12 (12.05) | 64.15 (11.71) | 63.13 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 8 | 15 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Duration of diabetes [Mean (Standard Deviation); unit: years] — Duration of diabetes mellitus in years
  years | 16.08 (8.52) | 21.3 (9.57) | 18.5 (9.3)
Arterial hypertension [Count of Participants; unit: Participants] | 26 | 24 | 50
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 136.68 (25.07) | 140.86 (26.29) | 138.77 (25.68)
Level of education [Count of Participants; unit: Participants]
  Incompleted elementary school | 14 | 10 | 24
  Completed elementary school | 4 | 7 | 11
  Incompleted high school | 6 | 6 | 12
  High school or more | 2 | 4 | 6
Access to smartphone [Count of Participants; unit: Participants] | 26 | 26 | 52
Access to computer [Count of Participants; unit: Participants] | 8 | 7 | 15
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of Hemoglobin A1c] — The HbA1c test result is delivered as a percentage. The higher the percentage, the higher the blood glucose level. Population: Only participants who completed the intervention
  percentage of Hemoglobin A1c
    number analyzed (Participants) | 19 | 12 | 31
    (all) | 8.2 (2.23) | 7.37 (1.41) | 7.86 (1.82)
Glycemic control [Count of Participants; unit: Participants] — glycemic control is considered when HbA1c is ≤ 8.0 %
  Participants | 14 | 20 | 34
Glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73 m^2] — Population: Participants who completed the intervention
  ml/min/1.73 m^2
    number analyzed (Participants) | 19 | 12 | 31
    (all) | 32.66 (12.28) | 28.28 (10.56) | 30.97 (11.42)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Determination of glycated hemoglobin (HbA1c) levels at the beginning and end of the nutritional intervention through teleconsultation and face-to-face consultation offered monthly for 4 months.
Time Frame: Baseline and at 4 month
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Teleconsultation | Face-to-face Consultation
Number analyzed (Participants) | 19 | 12
percentage of HbA1c | 7.4 (1.83) | 7.35 (2.25)
Statistical Analysis 1: Comparison: Teleconsultation vs Face-to-face Consultation; U Mann Whitney was used for inter-group comparison; Test type: Superiority; p = 0.37, t-test, 2 sided — The threshoid for statistical significance was p <0.05; Mean Difference (Final Values) = -1.76, Standard Deviation 0.8

2. Primary Outcome: Renal Function
Description: Determination of the estimated glomerular filtration rate (eGFR), at the end of the nutritional intervention through teleconsultation and face-to-face consultation offered monthly for 4 months.
Time Frame: Baseline and at 4 month
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Arm/Group | Teleconsultation | Face-to-face Consultation
Number analyzed (Participants) | 19 | 12
ml/min/1.73 m^2 | 34.45 (14.7) | 36.19 (27.61)
Statistical Analysis 1: Comparison: Teleconsultation vs Face-to-face Consultation; Test type: Superiority; p = 0.46, t-test, 2 sided — The threshold for statistical significance was p<0.05; U Mann Whitney was used for inter-group comparison; Mean Difference (Final Values) = -1.76, Standard Deviation 0.8

3. Secondary Outcome: Number of Participants With Adherence to Treatment
Description: To know the adherence to the level of compliance was assessed using a self-reported Likert scale in both study groups. Being the score 10 = good adherence and the score 1 = poor adherence to treatment.
Time Frame: Baseline and at 5 month
Measure: Count of Participants; unit: Participants
Arm/Group | Teleconsultation | Face-to-face Consultation
Number analyzed (Participants) | 19 | 12
Participants
  5 to 6 Likert scale | 0 | 2
  7 to 8 Likert scale | 15 | 7
  9 to 10 Likert scale | 4 | 3
Statistical Analysis 1: Comparison: Teleconsultation vs Face-to-face Consultation; Test type: Superiority; p = 0.16, Chi-squared

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Teleconsultation | Face-to-face Consultation
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/12
Other Adverse Events (participants affected / at risk) | 0/19 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teleconsultation (N=19) | Face-to-face Consultation (N=12)
Cancer (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03344549/Prot_SAP_ICF_000.pdf